CLINICAL TRIAL: NCT02231879
Title: A Phase III Double-Blind Randomized Crossover Study of Plerixafor Versus G-CSF in the Treatment of Patients With WHIM Syndrome.
Brief Title: Plerixafor Versus G-CSF in the Treatment of People With WHIM Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 140185; 14-I-0185 (Other: NIHCC)
Record Dates: First submitted 2014-09-03; First posted 2014-09-04 (Estimated); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2021-03

CONDITIONS: Myelokathexis; Infections; Neutropenia; Warts; Hypogammaglobulinemia
Keywords: Immunodeficiency; Neutropenia; Mozobil; Myelokathexis; Warts
MeSH Terms: conditions — Infections; Neutropenia; Warts; Agammaglobulinemia; Immunologic Deficiency Syndromes | interventions — plerixafor; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Plerixafor first then G-CSF (PG) (Active Comparator): Study drugs were both given subcutaneously twice daily for 14 months using unmarked prefilled glass syringes
  Interventions: Drug: Plerixafor; Drug: G-CSF
- G-CSF first then Plerixafor (GP) (Active Comparator): Study drugs were both given subcutaneously twice daily for 14 months using unmarked prefilled glass syringes
  Interventions: Drug: Plerixafor; Drug: G-CSF

INTERVENTIONS:
Drug: Plerixafor — Twice daily low dose injection for 14 months.
  Other Names: Mozobil
Drug: G-CSF — Twice daily low dose injection for 14 months.
  Other Names: Neupogen

SUMMARY:
Background:

- WHIMS (Warts, Hypogammaglobulinemia, Infections, and Myelokathexis Syndrome) is a rare disease. It can cause cancers, infections, and warts. Researchers want to see if a drug called plerixafor can treat WHIMS.

Objective:

- To compare plerixafor versus granulocyte colony stimulating factor (G-CSF) for preventing infections in people with WHIMS.

Eligibility:

- People ages 10-75 with WHIMS who have a CXCR4 gene mutation.

Design:

* Participants will be screened with a medical history, physical exam, and blood and urine tests. They may have heart and spleen tests and body scans. They may have samples of skin or warts taken. Researchers may take photographs of warts.
* Participants will start twice daily self-injections of G-CSF. Their doctors will decide the dosage.
* Initial Period (4-12 weeks)
* Participants will:
* continue the injections and their usual antibiotics and/or immunoglobulin
* have blood drawn
* keep a daily health diary
* Participants will visit the clinic for 2 days without injections.
* Adjustment Period 1 (8 weeks):
* Participants will:
* continue twice daily injections from home
* continue the daily health diary
* have blood tests every 2 weeks.
* Treatment Year 1:
* Participants will
* receive either plerixafor or G-CSF injections twice daily
* continue the health diary
* have blood tests every 2 months
* visit the clinic about every 4 months
* At the end of year 1, participants will visit the clinic for an evaluation. They will switch to the other study drug. They will have an 8-week adjustment and 1-year treatment period.
* At the end of year 2, participants will visit the clinic to complete their injections and go back to their previous G-CSF regimen. Participants will continue their daily health diary and have blood tests for 5-6 months.

DETAILED DESCRIPTION:
Warts, hypogammaglobulinemia, infections, and myelokathexis syndrome (WHIMS) is a rare combined primary immunodeficiency disorder caused by gain-of-function mutations in the gene for the chemokine receptor CXCR4. Normally, CXCR4 is expressed on most leukocyte subsets and functions in part to promote hematopoietic stem cell (HSC) and neutrophil homing to and retention in bone marrow. WHIM mutations alter the CXCR4 carboxyl terminus, which enhances and prolongs receptor signaling. As a result, egress of normally produced and functional neutrophils from the bone marrow to the blood is impaired causing neutropenia, a bone marrow pathologic finding referred to as myelokathexis. A similar mechanism may also affect other leukocyte subsets since WHIM patients usually are panleukopenic. Consequently, WHIM patients are predisposed to frequent acute bacterial infections, especially in the sinopulmonary tract, that may cause chronic morbidity, respiratory insufficiency and in some cases premature death. WHIM patients also have marked difficulty clearing infections with Human Papillomavirus (HPV), resulting in persistent cutaneous and anogenital warts that in several reported cases have evolved into cancer. Several deaths have also occurred due to cancer associated with Epstein -Barr virus (EBV) infection. Therapies currently used for WHIMS are non-specific and expensive, and include Granulocyte Colony-Stimulating Factor (G-CSF) (the drug currently approved by the Food and Drug Administration (FDA) to treat severe congenital neutropenia), intravenous immunoglobulin (IVIg), and prophylactic antibiotics. None of these measures has been formally evaluated for efficacy in WHIM syndrome (WHIMS); however, in our clinical experience based on the treatment of 24 WHIM patients seen at the National Institutes of Health (NIH) since 2006, recurrent bacterial infections continue to occur, despite the fact that the absolute neutrophil count (ANC) can be readily maintained above 500 cells/microliter by G-CSF and IgG levels can be restored to the normal range by IVIg. Thus, there continues to be a major unmet medical need for effective therapy in WHIMS despite the availability and application of best therapy for neutropenia and hypogammaglobulinemia in these patients. Plerixafor (Mozobil ) is a specific small molecule antagonist of CXCR4, licensed by the FDA for HSC mobilization for transplantation in cancer, and is therefore a logical candidate for molecularly targeted treatment of WHIMS. The goal of treatment would be to reduce CXCR4 signaling to normal, not to zero, thus, absent any off-target effects, targeted chronic treatment with this agent may be safe. In this regard, 2 recent short term Phase I dose-escalation studies of plerixafor, one from our group, in a total of 9 patients demonstrated that the drug could safely mobilize not only neutrophils, but also all other leukocyte subsets that are decreased in the blood of WHIM patients. A follow-up Phase I study, conducted by our group, in 3 patients given plerixafor 0.02-0.04 mg/kg/d for 6 months demonstrated that these hematopoietic effects were durable. Moreover, the frequency of infection was reduced on plerixafor as compared to retrospective data mined for the three years before starting therapy and prospective data collected for one year after ending therapy, even though 2 of the patients were taking GCSF during the comparison time periods. No new warts occurred during treatment and several existing warts improved or resolved. Although these results are encouraging, the small number of patients studied, limited duration of drug treatment, and retrospective mining of control data leave open to question whether plerixafor is truly efficacious for clinical outcomes in WHIMS. The randomized, double blinded, crossover trial described here is designed to answer this question by establishing the long-term safety and clinical efficacy (primary endpoint: infection severity; multiple secondary endpoints including wart control) of plerixafor as compared to G-CSF in the treatment of WHIMS patients 10-75 years of age. G-CSF as a comparator is required because of its approved use in patients with severe congenital neutropenia (SCN).

Brief outline of study we intend to randomize 20 patients and treat them in a double-blinded manner for 1 year with G-CSF and 1 year with plerixafor using a crossover design to allow direct comparison of infection severity during treatment with both agents, at doses determined by the patient s individual neutrophil response. A schedule of events has been provided in Appendix A. Data will be analyzed as specified in the Statistics section (Section 14) after randomization. Tolerability and patient drug preference will also be assessed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects are eligible to enter the study if they meet all of the following criteria:

1. Age greater than or equal to 10 and less than or equal to 75 years.
2. Heterozygous mutation in the C-tail of CXCR4 in addition to a clinical diagnosis of WHIMS.
3. Documented neutropenia with a baseline ANC below 1500 cells/microL of blood.
4. History of severe and/or recurrent infections.
5. Willingness to interrupt G-CSF medication, 2 days prior to study drug injection.
6. Must have a local medical provider for medical management.
7. Must be willing to provide blood, plasma, serum, and DNA samples for storage.
8. All study subjects must agree not to become pregnant or impregnate a female. Women of childbearing potential must agree to take appropriate steps to avoid becoming pregnant for the duration of the study. Participants in whom pregnancy is biologically possible must use at least 2 study approved methods of contraception, one of which must be a barrier method, and must continue contraception until 5 months after stopping the study drug:

   * Male or female condoms with a spermicide,
   * Diaphragm or cervical cap with spermicide,
   * Intrauterine device,
   * Contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive,
   * Male partner with vasectomy and documented aspermatogenic sterility.
9. Willingness to comply with the study medications, visits, and procedures, as deemed necessary by the principal investigator (PI).

EXCLUSION CRITERIA:

If any of the following exclusion criteria are met, a subject will not be enrolled in this study:

1. Neutropenia due to maturation defects in the myeloid lineage or a type of neutropenia, which in the investigator s opinion, is unlikely to improve from the medication administered in this study.
2. Pregnant or breast-feeding women.
3. Known hypersensitivity to plerixafor, G-CSF, or any components of the products.
4. Predisposition to or history of life-threatening cardiac arrhythmia.
5. Requiring dialysis or having markedly impaired renal function with a Creatinine Clearance (CrCl) <15 mL/min.
6. Condition that in the investigator s opinion places a subject at undue risk by participating in the study.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H McDermott, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDermott DH, Velez D, Cho E, Cowen EW, DiGiovanna JJ, Pastrana DV, Buck CB, Calvo KR, Gardner PJ, Rosenzweig SD, Stratton P, Merideth MA, Kim HJ, Brewer C, Katz JD, Kuhns DB, Malech HL, Follmann D, Fay MP, Murphy PM. A phase III randomized crossover trial of plerixafor versus G-CSF for treatment of WHIM syndrome. J Clin Invest. 2023 Oct 2;133(19):e164918. doi: 10.1172/JCI164918. PMID 37561579
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-I-0185.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 subject could not tolerate minimal possible dose of G-CSF (Neupogen) 15 micrograms subcutaneously twice daily during screening period and was not randomized
Groups:
- Plerixafor First Then Filgrastim; Filgrastim First Then Plerixafor: G-CSF or plerixafor, blinded
  Plerixafor: Twice daily low dose injection for 14 months.
  G-CSF: Twice daily low dose injection for 14 months.
Period: Overall Study
Arm/Group | Plerixafor First Then Filgrastim | Filgrastim First Then Plerixafor
Started | 10 | 9
Completed | 8 | 7
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plerixafor First Then Filgrastim | Filgrastim First Then Plerixafor | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 4 | 5
  Between 18 and 65 years | 9 | 5 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15
  El Salvador | 1 | 0 | 1
  Sweden | 1 | 0 | 1
  Spain | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Severity of Infection
Description: The primary outcome is a Total Infection Severity Score (TISS). Each infection during the 12 month period of treatment on each drug was scored for severity on a scale of 1-10 with higher scores representing more severe infections and then these scores were summed (weighted based on time at risk) to create a total infection severity score (TISS) in each period for each participant (range 0 to infinity). Drug failures during a period were pre-defined to count as more extreme than any TISS score. The primary analysis outcome is based on the Difference in Total Infection Severity Score (TISS) in Period 1 minus TISS in Period 2 analysis, with drug failures in only one period assigned the highest absolute value for the difference, with the sign defined according to the treatment order (e.g., negative for period 2 drug failures only). Higher values of the difference represent a worse outcome in the first period than in the second period. Thus, each participant's infection severity
Time Frame: Scores from 12 months treatment on each study drug
Population: There are 19 participants that started both periods, 1 participant had drug failure during both periods, 3 participants had drug failure only during the period on Plerixafor. The outcome measure data table only summarizes the periods that were not drug failures, but the primary analysis includes the treatment failure periods by giving them the most extreme score (see Statistical Analysis section).
Measure: Median (Full Range); unit: score on a scale (with no maximum)
Groups:
- G-CSF (Both Periods Combined): This group of observations are the outcomes (TISS=total infection severity score) during the period when each participant received G-CSF (i.e., filgrastim). Since each participant had one period on G-CSF, we have outcomes on all participants that started in participant flow, except those that had treatment failure.
  Recall, this is a crossover trial, where participants were randomized to receive either (PG) Plerixafor in Period 1 then G-CSF (i.e., filgrastim) ( in Period 2 or (GP) G-CSF in Period 1 then Plerixafor in Period 2. For example participants randomized to PG were given plerixafor twice daily subcutaneously for a total of 14 months (2 months dose adjustment followed by 12 months of treatment where infections and other parameters were evaluated) then crossover occurred and G-CSF was given twice daily subcutaneously over a total of 14 months (2 months dose adjustment followed by 12 months of treatment where infections and other parameters were evaluated).
- Plerixafor (Both Periods Combined): This group of observations are the outcomes (TISS=total infection severity score) during the period when each participant received Plerixafor. Since each participant had one period on Plerixafor, we have outcomes on all participants that started in participant flow, except those that had treatment failure.
  Recall, this is a crossover trial, where participants were randomized to receive either (PG) Plerixafor in Period 1 then G-CSF (i.e., filgrastim) ( in Period 2 or (GP) G-CSF in Period 1 then Plerixafor in Period 2. For example participants randomized to PG were given plerixafor twice daily subcutaneously for a total of 14 months (2 months dose adjustment followed by 12 months of treatment where infections and other parameters were evaluated) then crossover occurred and G-CSF was given twice daily subcutaneously over a total of 14 months (2 months dose adjustment followed by 12 months of treatment where infections and other parameters were evaluated).
Arm/Group | G-CSF (Both Periods Combined) | Plerixafor (Both Periods Combined)
Number analyzed (Participants) | 18 | 15
score on a scale (with no maximum) | 12.5 [0 to 36] | 9 [0 to 24]

2. Primary Outcome: Difference in Total Infection Severity Score
Description: The primary outcome is a difference: the Total Infection Severity Score (TISS) in Period 1 minus the TISS in Period 2. Higher values represent a worse outcome in the first period than in the second period. Each infection during the 12 month period of treatment on each drug was scored for severity on a scale of 1-10 with higher scores representing more severe infections and then these individual infection scores were summed (weighted by time at risk) to create a total infection severity score (TISS) in each period. Because there is no pre-determined number of infections, the range is -infinity to +infinity. If a participant has a drug failure in only one period, their difference rank is either the highest rank (if the failure is in Period 1) or the lowest rank (if the failure is in Period 2), failure on both periods gives a difference of 0. 1 subject failed on both treatments, and 3 subjects failed only on plerixafor.
Time Frame: Scores from 12 months treatment on each study drug
Population: The two populations are the two randomization arms in the crossover trial.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Plerixafor in Period 1 and G-CSF in Period 2: Participants were given plerixafor twice daily subcutaneously for a total of 14 months (2 months dose adjustment followed by 12 months of treatment where infections and other parameters were evaluated) then crossover occurred and G-CSF was given twice daily subcutaneously over a total of 14 months (2 months dose adjustment followed by 12 months of treatment where infections and other parameters were evaluated).
- G-CSF in Period 1 and Plerixafor in Period 2: Participants were given G-CSF twice daily subcutaneously for a total of 14 months (2 months dose adjustment followed by 12 months of treatment where infections and other parameters were evaluated) then crossover occurred and Plerixafor was given twice daily subcutaneously over a total of 14 months (2 months dose adjustment followed by 12 months of treatment where infections and other parameters were evaluated).
Arm/Group | Plerixafor in Period 1 and G-CSF in Period 2 | G-CSF in Period 1 and Plerixafor in Period 2
Number analyzed (Participants) | 10 | 9
score on a scale | 10.6 [1 to 19] | 9.33 [1 to 19]
Statistical Analysis 1: Comparison: Plerixafor in Period 1 and G-CSF in Period 2 vs G-CSF in Period 1 and Plerixafor in Period 2; This was a pre-specified primary analysis plan, and the two arms are compared with a Wilcoxon-Mann-Whitney test on the primary outcome. This is non-standard (since both arms contain both treatment groups), however, it is a valid test by randomization since it is a permutation test. The statistic of TISS in Period 1 minus TISS in Period 2 was chosen so that even if there are carry-over effects this will give a valid test; Test type: Superiority — This is a two-sided test, with the null hypothesis that the distribution of the difference scores is the same in both arms; p = 0.65, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons, since this is the only pre-specified primary analysis. P<=0.05 is considered significant
Statistical Analysis 2: Comparison: Plerixafor in Period 1 and G-CSF in Period 2 vs G-CSF in Period 1 and Plerixafor in Period 2; Maintenance of absolute lymphocyte count greater than 1000 cells/microliter measured 3 hours after a dose for plerixafor as compared to G-CSF; Test type: Superiority; p < 0.0001, McNemar — Not adjusted for multiple comparisons, one-sided test, a priori significance set at 0.025
Statistical Analysis 3: Comparison: Plerixafor in Period 1 and G-CSF in Period 2 vs G-CSF in Period 1 and Plerixafor in Period 2; Maintenance of absolute neutrophil counts >500 cells/microliter for G-CSF versus plerixafor measured as the proportion of successes (75% of measured) while on G-CSF minus the proportion on plerixafor; Test type: Non-Inferiority — Pre-specified non-inferiority margin of 0.40 which was estimated to be about 50% of the effect size of G-CSF versus placebo; p = 0.023, McNemar — Not adjusted for multiple comparisons, one-sided test, a priori significance set at 0.025

ADVERSE EVENTS:
Time Frame: up to 14 months on each study drug
Description: Definitions were identical to those as listed on clinicaltrials.gov. Adverse events were obtained from repeated in-person participant evaluation approximately every 4 months and laboratory testing approximately every 2 months during each drug treatment.
Arm/Group | G-CSF | Plerixafor
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 6/19 | 2/19
Other Adverse Events (participants affected / at risk) | 19/19 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-CSF (N=19) | Plerixafor (N=19)
Flu-like illness (Infections and infestations) | 1 (1) | 0 (0) — Dehydration requiring intravenous fluids
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Probable Reactive
pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) — hospitalized
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-CSF (N=19) | Plerixafor (N=19)
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 1 (3) | 1 (2)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (13) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Acute bronchitis (Infections and infestations) | 9 (19) | 2 (7)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (8) | 6 (11)
Upper respiratory infection (Infections and infestations) | 2 (5) | 3 (7)
Otitis media (Infections and infestations) | 6 (8) | 1 (4)
Gastroenteritis (Infections and infestations) | 6 (8) | 0 (0)
Herpes simplex (Infections and infestations) | 3 (5) | 2 (3)
Urinary Tract Infection (Infections and infestations) | 4 (6) | 2 (2)
Acute sinusitis (Infections and infestations) | 4 (5) | 2 (2)
Abscess (Infections and infestations) | 2 (4) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (3) | 2 (2)
Pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Skin Infection (Infections and infestations) | 2 (2) | 1 (1)
Tinea capitis (Infections and infestations) | 1 (1) | 1 (2)
Conjunctivitis (Infections and infestations) | 2 (3) | 0 (0)
Infectious Diarrhea (Infections and infestations) | 1 (2) | 1 (1)
Tinea corporis (Infections and infestations) | 0 (0) | 2 (2)
Herpes labialis (Infections and infestations) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ankle sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (5) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 3 (4)
Weight gain (Investigations) | 2 (2) | 5 (5)
Creatinine increased (Investigations) | 2 (2) | 2 (2)
Bone mineral content decreased (Investigations) | 2 (2) | 1 (1)
CPK increased (Investigations) | 2 (2) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (6) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 14 (41) | 7 (7)
Knee pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (7) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4)
Low back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 6 (12) | 3 (5)
Migraine (Nervous system disorders) | 1 (1) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 3 (11) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Papular rash (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Pruritic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Elective surgery (Surgical and medical procedures) | 2 (4) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
1. Highly variable disease phenotypic expression made crossover design optimal but a placebo arm was not included due to infection risk of severe neutropenia
2. Prophylactic supplemental immunoglobulin and antibiotics were allowed
3. Tolerance of G-CSF was insured prior to randomization but plerixafor was never used before randomization in 17/19 patients,
4. Non-inferiority analysis of primary endpoint was not planned because there were no defined equivalence margins

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT02231879/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT02231879/ICF_001.pdf